CLINICAL TRIAL: NCT01474707
Title: Assessing Chronic Obstructive Pulmonary Disease (COPD) Knowledge, Beliefs, and Health Literacy in Chinese Immigrant Adults With a Diagnosis of COPD
Brief Title: Educational Interventions for Chronic Obstructive Pulmonary Disease (COPD) Self-management in Ethno-cultural Communities
Acronym: COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Vancouver Coastal Health (Other Government); Main Line Health (Other); Provincial Health Services Authority British Columbia (Other); Vancouver Foundation (Other); Heart and Stroke Foundation of Canada (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Mark Fitzgerald, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H09-02069
Record Dates: First submitted 2011-11-03; First posted 2011-11-18 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; Educational materials; Cultural background; Instructional videos; Patient education handouts; Lung age
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — One-Carbon Group Transferases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group one (Experimental): Group1 will view the knowledge-based video only
  Interventions: Behavioral: Group one
- Group two (Experimental): Group two will view the motivational video only
  Interventions: Behavioral: Group two
- Group three (Experimental): Group three will view both knowledge-based and motivational videos
  Interventions: Behavioral: Group three
- Group four (Experimental): Group four will view the printed educational pamphlet and will not view either video
  Interventions: Behavioral: Group four

INTERVENTIONS:
Behavioral: Group one — Group 1 will view the knowledge-based video only
  Arms: Group one
Behavioral: Group two — Group two will view the motivational video only
  Arms: Group two
Behavioral: Group three — Group three will view both knowledge-based and motivational videos
  Arms: Group three
Behavioral: Group four — Group four will view the printed educational pamphlet and will not view either video
  Arms: Group four

SUMMARY:
Goal: The main goal of this study is to develop and validate educational materials that aim to improve self-management knowledge and practices about COPD among patients in Mandarin and Cantonese-speaking communities in the Greater Vancouver Area (GVA).

Objectives: "1." To assess the current landscape of COPD beliefs, perceptions and practices, as well as health literacy as it relates to Chinese Mandarin and Cantonese-speaking patients; "2." To develop effective partnerships within primary care physicians serving Chinese newcomers in the GVA' "3." To conduct focus group sessions with collaborative primary care physicians to identify common factors that contribute to under service and access barriers among patients in the target communities; "4." To assess the effectiveness of the educational materials on patients' beliefs, perceptions, practices, and health literacy related to COPD control and self-management; and "5." To improve the capacity of physicians and allied health workers in primary care settings in educating patients and their families about self-management of COPD.

The implementation of the project will include the following phases: "1." Build and strengthen established partnerships with primary care practices serving newcomers in GVA; "2." Conduct an environmental scan and needs assessment (literature review, interviews and focus groups with community members and key-informants); "3." Development of story scripts, video clips and other educational materials, and relevant measurement tools; "4." Application of the video clips and other educational materials to test their effectiveness on health literacy, beliefs, and knowledge among COPD patients from the target communities; and "5." Evaluation of the usefulness of videos and other educational materials, and the project's process and outcomes.

DETAILED DESCRIPTION:
The main aim of this project is to address our knowledge gap about COPD management, access problems, and differences in environmental exposure among newcomers in Canada: by engaging key stakeholders, fostering dialogue, gathering baseline data, and generating knowledge on how improved access to culturally and linguistically appropriate educational materials can enhance awareness and practices about COPD control and self-management through interventional study, thereby improving the health status of the target populations. We plan to document: "1." what are the cultural imperatives that are likely to mediate ethnic Chinese patients to manage COPD? "2." to what extent does the Canadian health care system's environment influence newcomers response to COPD? Our aim is to examine the belief system and health practices among target communities that may influence treatment and management of COPD.

This research will make theoretical, methodological and applied research contributions. It will establish strong community - primary care provider and academic connections for the development of the proposed educational materials, measurement tools, and framework. Community participation will be included throughout the development of this study, enhancing the potential of acquiring new knowledge about cultural and traditional practices of the sample population.

Our approach will enable primary health care providers, knowledge users, and policy makers to design appropriate educational intervention initiatives targeted to diverse ethnic minority groups in relation to COPD. We foresee findings that provide not only better ways to measure health literacy pertaining to COPD in our target populations, but that will also help develop materials and measures that can be applied to other populations in BC and the rest of Canada. We expect that the participatory approach used in this study will contribute to capacity building, improving newcomers' ability to access and use relevant COPD information (in terms of prevention, control and management) and to transfer and share the information learned with other members of the target communities. The proposed community consultation will also help us identify culturally appropriate communication mode(s) to deliver health information messages and determine practical adult learning approaches applicable to diverse communities in Canada.

ELIGIBILITY:
Inclusion Criteria:

* A physician diagnosed COPD patients
* Be at least 21 years old
* Speaks Mandarin or Cantonese
* Immigrated to Canada in the past 15 years from mainland China or Hong Kong

Exclusion Criteria:

* Self-reported patients
* Person under 21 years old
* Person who lives in a nursing home
* Unwilling to participate in the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-01; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Using study questionnaire to measure knowledge about COPD control and self-management | Six months
  The investigators will assess participants knowledge about COPD management and control at initial visit (baseline), and will then assess it again two more times: at month two (post-test) and month six (follow-up post-test). The investigators will then compare the changes in the participants' knowledge within this six-month period; from initial visit to follow-up post-test.

SECONDARY OUTCOMES:
Assessing the target community cultural beliefs and practices and systemic barriers that are likely interfere Chinese patients to manage their COPD | Four months
  The investigators will conduct two focus group sessions (one in Mandarin and one in Cantonese) with Chinese key-informants, COPD patients, primary care partners, and members of the study Community Advisory Committee to discuss and brainstorm about the cultural, language, and systemic barriers that prevent patient from Chinese community to self-manage their COPD.
Educational materials development | Four months
  The investigators will develop educational materials for this study (including video clips and patient handouts) through a participatory action approach with direct involvement of Chinese key informants, media people, study collaborators, and community members. The investigators will develop two motivational and two knowledge-based videos, as well as two pictorial pamphlets.

CONTACTS AND LOCATIONS:
Overall Officials: Mark J FitzGerald, M.D., Principal Investigator — University of British Columbia
Locations (2):
- Canada (2):
  - Centre for Clinical Epidemiology and Evaluation, Vancouver Coastal Health Research Institute, Vancouver, British Columbia
  - University of British Columbia - Vancouver Coastal Health, Vancouver, British Columbia

REFERENCES:
- [Result] Poureslami I, Kwan S, Lam S, Khan NA, FitzGerald JM. Assessing the effect of culturally specific audiovisual educational interventions on attaining self-management skills for chronic obstructive pulmonary disease in Mandarin- and Cantonese-speaking patients: a randomized controlled trial. Int J Chron Obstruct Pulmon Dis. 2016 Aug 3;11:1811-22. doi: 10.2147/COPD.S105408. eCollection 2016. PMID 27536093
- See also: UBC Lung Centre — http://www.thelungcentre.ca
- See also: UBC Institute for Heart and Lung Health — http://heartandlung.ca/